CLINICAL TRIAL: NCT05187325
Title: The Effect of Myofascial Trigger Points on Clinical Symptoms, Pain and Limitation of Temporomandibular Joint Function in Disc Displacement With Reduction
Brief Title: The Clinical Effects of Myofascial Trigger Points in Disc Replacement With Reduction
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Merve Damla Korkmaz, Specialist Doctor, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: KAEK/2021.11.309
Record Dates: First submitted 2021-12-25; First posted 2022-01-11 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Temporomandibular Joint Disorders; Myofascial Trigger Point Pain; Jaw Diseases; Pain
Keywords: temporomandibular joint; disc displacement with reduction; trigger point; pain level
MeSH Terms: conditions — Temporomandibular Joint Disorders; Myofascial Pain Syndromes; Jaw Diseases; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- myofascial trigger point and disc displacement with reduction: the participants have myofascial trigger points in master muscle and also temporomandibular joint disc displacement with reduction.
  Interventions: Other: no intervention
- disc displacement with reduction: the participants have only temporomandibular joint disc displacement with reduction.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — there is no intervention

SUMMARY:
This is a prospective, and controlled trial. 60 participants with myofascial trigger points and disc displacement with reduction and 60 participants with disc displacement with reduction will be included in the study. These two groups will be compared for clinical findings, pain severity and limitation of the temporomadibular function.

DETAILED DESCRIPTION:
This is a prospective, and controlled trial. 60 participants with myofascial trigger points and disc displacement with reduction and 60 participants with disc displacement with reduction will be included in the study. The participants' ages will be between 18-65 years of both genders.

These two groups will be compared for clinical findings with DC/TMD Axis I- Symptom Questionnaire, pain levels in the last 1 month with DC/TMD Axis II-Graded Chronic Pain Scale, and limitation of the temporomadibular function with DC/TMD Axis II-Jaw Functional Limitation Scale-8.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old of both genders.
* Presence of disc displacement with reduction with/without myofascial trigger points in master muscles.
* Being accepted of the participation in the study.

Exclusion Criteria:

* Lack of cognitive ability to understand test instructions, illiteracy, aphasia, presence of a known psychiatric illness
* Refusal to participate in the study
* Patients under the age of 18 and over the age of 65
* Having other temporomandibular joint disorders other than the diagnosis of RDD and/or myofascial trigger points

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants who ages between 18-65 years of both genders with disc displacement with reduction with/ without myofascial trigger points in master muscles will be included in the study.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
mouth opening distance | 1 day
  Maximal opening of mouth is described as the greatest distance between incisal edge of maxillary central incisor to the incisal edge of mandibular central incisor, when the mouth is opened as wide as possible painlessly or as the inter incisal distance plus the overbite.
bruxism | 1 day
  bruxism is a stereotyped movement disorder characterized by grinding or clenching of the teeth
limitation of the movement of the temporomandibular joint | 1 day
  limitation of the movement of the temporomandibular joint
temporomandibular joint noises | 1 day
  noises of the temporomandibular joint
locking of the temporomandibular joint | 1 day
  locking of the temporomandibular joint
Graded Chronic pain Scale v.2.0 | 1 day
  Version 2 of the GCPS includes, in addition to the 3 items for pain intensity and 4 items for function, one item for number of days of pain.
Jaw Functional Limitation Scale-8 | 1 day
  The JFLS was initially developed as an 8-item global scale for overall functional limitation of the masticatory system; based on the resultant items and supporting psychometric data, the instrument was re-developed in order to expand measured constructs to also include masticatory limitation, vertical mobility limitation, and verbal and non-verbal communication limitation.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Kucukcekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
It will be decided after the publication